CLINICAL TRIAL: NCT05053542
Title: The Necessity of Preoperative Bowel Preparation for Hemorrhoidectomy: A Single-Center Retrospective Comparative Study
Brief Title: The Necessity of Preoperative Bowel Preparation
Status: Completed | Type: Observational
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: N202009024
Record Dates: First submitted 2021-08-30; First posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-08

CONDITIONS: Pain, Postoperative; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Enema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- With or without enema before operation: Patients who had received pre-operative bowel preparation(PBP) were identified using electronic medical records. Patients prescribed an enema solution (EVAC enema 118 mL/bot, Purzer Pharmaceutical Co., Ltd) before surgery were allocated to the PBP group. Patients who received no PBP were allocated to none PBP group.
  Interventions: Procedure: Enema

INTERVENTIONS:
Procedure: Enema — Patients in the PBP group underwent a cleansing enema procedure with a solution of monosodium phosphate and disodium phosphate (EVAC enema 118 mL/bot, Purzer Pharmaceutical Co., Ltd) before hemorrhoidectomy, whereas patients in the non-PBP group skipped the procedure.

SUMMARY:
Hemorrhoidectomy is an common treatment for high-grade hemorrhoids. The necessity of preoperative bowel preparation (PBP) in hemorrhoidectomy is inconclusive. This study aims to evaluate the benefit and safety of PBP in hemorrhoidectomy.

DETAILED DESCRIPTION:
Hemorrhoidectomy is an effective treatment for high-grade hemorrhoids and is recommended in patients with grade III-IV hemorrhoids. Common hemorrhoidectomy approaches include stapled hemorrhoidopexy and conventional procedures, such as Ferguson hemorrhoidectomy and Milligan-Morgan hemorrhoidectomy. Conventional techniques produce a lower recurrence rate, whereas stapled hemorrhoidopexy is associated with fewer postoperative complications and shorter recovery time.

Common complications after hemorrhoidectomy include urinary retention, pain, and delayed hemorrhage. Surgical site infection is a rare complication after hemorrhoid excision. Traditional opinions held that preoperative bowel preparation (PBP) reduces fecal mass and bacterial count in the bowel lumen, minimizing the risk of infective and anastomotic complications. However, a study that evaluated intramucosal bacterial count demonstrated that PBP does not reduce the colon bacterial count. A randomized control trial (RCT) evaluating the effect of PBP before colorectal surgery suggested that the procedure can be omitted. However, another RCT with 79 participants revealed that bowel preparation before anorectal surgery can result in less pain during the first postoperative defecation. A meta-analysis with 36 studies concluded that PBP before elective colorectal surgery does not affect the postoperative complication rate. On the contrary, the necessity of PBP before anorectal surgeries remains unreported. The choice of whether PBP has to be performed is often the surgeon's preference. It may be challenging for physicians to determine the appropriate decision of PBP before hemorrhoidectomy to reduce postoperative complications while minimizing patient discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent hemorrhoidectomy

Exclusion Criteria:

* Patients who had received emergent or other anorectal surgery, such as fistulectomy, were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient underwent hemorrhoidectomy in Taipei Medical University Shuang-Ho Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Post-operative pain and | 4 weeks
  A numerical rating scale (NRS) was used for measuring daily postoperative pain, where 0 represented no pain and 10 represented the worst pain ever experienced.
Post-operative oral analgesic use. | 4 weeks
  The daily dose of oral analgesics was recorded to represent patients' dependence on medicine for postoperative pain control.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Shuang-Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided